CLINICAL TRIAL: NCT02574156
Title: Control of Hyperglycemia After Cardiac Surgery: CHyCS Trial
Acronym: CHyCS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Finished
Sponsor: University of Sao Paulo (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Eduesley Santana Santos, RN, Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin; Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Group (Experimental): Patients randomized for Conventional Group will receive insulin infusion of regular insulin (100 UI) in 100 mL of saline in continuous infusion pump for maintenance of blood glucose between 140 mg/dl and 180 mg/dl.
  Interventions: Drug: Insulin
- Moderate Group (Experimental): Patients randomized for ModerateGroup will receive insulin infusion of regular insulin (100 UI) in 100 mL of saline in continuous infusion pump for maintenance of blood glucose between 100 mg/dl and 130 mg/dl.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — All patients will receive insulin. However, the infusion flow will be different according to the group.
  Other Names: Glycemic Control

SUMMARY:
The investigators aim to study the impact of a strategy of a intensive glycemic control in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Patients undergoing heart surgery at the Heart Institute (InCor) will be randomized and in accordance with a list of random numbers, generated by a computer program, are allocated in one of the treatment groups (conventional or intensive) when the blood glucose value recorded is greater than 200 mg/dl on two consecutive measures in an interval of 30 minutes.Conventional Group (GCon): patients randomized to the conventional group will receive insulin infusion in a dilution of 100 units of regular insulin in 100 ml of physiological solution (NaCl 0.9%) in continuous infusion pump for maintenance of blood glucose between 140 mg/dl and 180 mg/dl.

Group intensive (GInt): patients randomized to the intensive group will receive insulin infusion in a dilution of 100 units of regular insulin in 100 ml of physiological solution (NaCl 0.9%) in continuous infusion pump for maintenance of blood glucose between 90 mg/dl and 110 mg/dl.

The insulin dose adjustment will be based on measurements of arterial blood glucose undiluted, held at intervals of one to 4 hours with the use of a monitoring system of glucose and beta-blood ketone (Freestyle Precision Pro, Abbott). The dosage is adjusted according to an algorithm by a team of intensive care nurses, trained for this purpose and assisted by a study physician not involved in the clinical care of patients.

On admission, all patients will receive intravenous glucose solution continuously (200 to 300 g in 24 hours). As soon as possible, the patient will be nurtured according to the routine of Surgical ICU for nutrition in the postoperative period of cardiac surgery patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing heart surgery;
* Age greater than 18 years;
* Sign the informed consent form;
* Capillary blood glucose greater than 200mg/dL ICU admission

Exclusion Criteria:

* Admitted for surgical repair of congenital heart defects;
* Dialytic Chronic renal failure;
* Participation in other research protocol;
* Diagnosis of HIV/AIDS;
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Infection of surgical wound infection | 30 days
  The primary outcome measure will be assessed according to the American Society of Thoracic Surgeons guidelines

SECONDARY OUTCOMES:
Need for reoperation | 30 days
  This outcome measure will be assessed according to the American Society of Thoracic Surgeons guidelines
Acute renal injury (defined by the KDIGO classification) | 30 days
  This outcome measure will be assessed according to the KDIGO Criterion
Infection of the bloodstream | 90 days
Prolonged mechanical ventilation | 90 days
Need for transfusion of blood products | 90 days
Occurrences of hypoglycemia | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Eduesley Santana Santos, Ph.D, Principal Investigator — University of Sao Paulo
Locations (1):
- Eduesley Santana Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Macrae D, Grieve R, Allen E, Sadique Z, Morris K, Pappachan J, Parslow R, Tasker RC, Elbourne D; CHiP Investigators. A randomized trial of hyperglycemic control in pediatric intensive care. N Engl J Med. 2014 Jan 9;370(2):107-18. doi: 10.1056/NEJMoa1302564. PMID 24401049
- [Result] Yates AR, Dyke PC 2nd, Taeed R, Hoffman TM, Hayes J, Feltes TF, Cua CL. Hyperglycemia is a marker for poor outcome in the postoperative pediatric cardiac patient. Pediatr Crit Care Med. 2006 Jul;7(4):351-5. doi: 10.1097/01.PCC.0000227755.96700.98. PMID 16738506
- [Result] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Result] Brunkhorst FM, Engel C, Bloos F, Meier-Hellmann A, Ragaller M, Weiler N, Moerer O, Gruendling M, Oppert M, Grond S, Olthoff D, Jaschinski U, John S, Rossaint R, Welte T, Schaefer M, Kern P, Kuhnt E, Kiehntopf M, Hartog C, Natanson C, Loeffler M, Reinhart K; German Competence Network Sepsis (SepNet). Intensive insulin therapy and pentastarch resuscitation in severe sepsis. N Engl J Med. 2008 Jan 10;358(2):125-39. doi: 10.1056/NEJMoa070716. PMID 18184958
- [Result] Preiser JC, Devos P, Ruiz-Santana S, Melot C, Annane D, Groeneveld J, Iapichino G, Leverve X, Nitenberg G, Singer P, Wernerman J, Joannidis M, Stecher A, Chiolero R. A prospective randomised multi-centre controlled trial on tight glucose control by intensive insulin therapy in adult intensive care units: the Glucontrol study. Intensive Care Med. 2009 Oct;35(10):1738-48. doi: 10.1007/s00134-009-1585-2. Epub 2009 Jul 28. PMID 19636533
- [Result] Dandona P, Mohanty P, Chaudhuri A, Garg R, Aljada A. Insulin infusion in acute illness. J Clin Invest. 2005 Aug;115(8):2069-72. doi: 10.1172/JCI26045. PMID 16075050
- [Result] Boyle EM Jr, Pohlman TH, Johnson MC, Verrier ED. Endothelial cell injury in cardiovascular surgery: the systemic inflammatory response. Ann Thorac Surg. 1997 Jan;63(1):277-84. doi: 10.1016/s0003-4975(96)01061-2. PMID 8993292
- [Result] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 3--valve plus coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S43-62. doi: 10.1016/j.athoracsur.2009.05.055. PMID 19559824